CLINICAL TRIAL: NCT04713306
Title: Gender Differences in Diagnostic Tools, Medication, Time to Medication and Non-motor Symptoms in Parkinsonian Patients- a Swedish Register Study
Brief Title: Gender Differences in Parkinsonian Patients- a Swedish Register Study
Status: Completed | Type: Observational
Sponsor: Region Jönköping County (Other Government)
Collaborators: Jonkoping University (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: XXXXX
Record Dates: First submitted 2020-10-06; First posted 2021-01-19 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: NonMotorSymptoms, medication, National Registries
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants in the Swedish Neuro Register: Participants are patients with parkinsonian symptoms

SUMMARY:
BACKGROUND: The complex impact of gender has been studied in different perspectives of health and disease in the literature. However, few attempts have been made to compile data from systematic disease specific registrations Swedish National Quality Registers play an important role in collecting large amounts of diagnose specific data, symptoms, and treatments. The subset Parkinson Registry has been in use for more than 20 years and are represented in all counties and hospitals where neurological care is provided in Sweden and offer optimal conditions to describe gender specific differences in the use of diagnostic tools, lead times and symptom profiles.

DETAILED DESCRIPTION:
Aim: To study differences between gender in diagnostic tools, pharmacological interventions, and self-reported symptoms in Parkinson´s Disease (PD).

METHODS:

Data were extracted from the Swedish Neuro Registers, one of the Swedish National Quality Registers. A mix of urban and rural parts of the country were chosen and data were divided by gender. Self-reported first experienced PD related symptom was used to define the starting point when processing the data. Zero to three years from this point was defined as early symptoms and over three years as late symptoms.

CONCLUSION:

Differences between gender were seen in all chosen aspects, both diagnostically. Distinctions were also prominent in reported NonMotorSymptoms (NMS) profiles. These findings should be important to take into consideration for patients, professional staff, and caregivers in the daily work with gender mixed PD groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants registered in the Swedish Neuro Registers.
* Parkinson´s Disease
* Acceptance of extraction of data

Exclusion Criteria:

* non parkinsonian patients
* Participants in the Registries who have not given allowance of extraction of data.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — yes self-representation
Study Population: Cohorts from rural areas and larger cities of Southern Sweden with diagnosed parkinsonism.
Sampling Method: Probability Sample
Enrollment: 1217 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Differences between gender | 2006-2020
  investigations, medications,NonMotorSymptoms

CONTACTS AND LOCATIONS:
Overall Officials: Johan Lokk, PhD, Study Director — Karolinska Institutet
Locations (1):
- FUTURUM, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No